CLINICAL TRIAL: NCT05774691
Title: Routine Versus Selective Protamine Administration to Reduce Bleeding Complications After Transcatheter Aortic Valve Implantation
Brief Title: Routine Versus Selective Protamine Administration to Reduce Bleeding Complications After Transcatheter Aortic Valve Implantation (POPular ACE TAVI)
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: St. Antonius Hospital (Other)
Collaborators: St. Antonius Research Fund (Unknown)
Responsible Party: Principal Investigator, Jurriën M. ten Berg, MD, PhD, MD, PhD, St. Antonius Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2023-504205-36-00
Record Dates: First submitted 2023-03-03; First posted 2023-03-20 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Aortic Valve Stenosis
Keywords: TAVI; TAVR; Bleeding; Mortality; Allergy; Protamine
MeSH Terms: conditions — Aortic Valve Stenosis; Hemorrhage; Hypersensitivity | interventions — Protamines

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Routine protamine administration (Active Comparator): Routine protamine administration in a ratio of 1 IE per 1 IE of unfractionated heparin.
  Interventions: Drug: Protamine sulfate
- Selective protamine administration (Active Comparator): Selective protamine administration, in case of (threatening) bleeding.
  Interventions: Drug: Protamine sulfate

INTERVENTIONS:
Drug: Protamine sulfate — Routine protamine administration in a ratio of 1 IE per 1 IE of unfractionated heparin.
  Other Names: Routine heparin reversal
  Arms: Routine protamine administration
Drug: Protamine sulfate — Selective protamine administration, in case of (threatening) bleeding
  Other Names: Selective heparin reversal
  Arms: Selective protamine administration

SUMMARY:
Heparin reversal by protamine administration after transcatheter aortic valve implantation (TAVI) may reduce bleeding events. However, protamine can also cause life-threatening allergic reactions. High-quality evidence regarding the clinical safety and efficacy of routine protamine administration after TAVI is lacking.

The aim of this clinical trial is to determine if routine protamine administration, compared with selective protamine administration, reduces the risk of all-cause mortality or clinically relevant bleeding within 30 days after transcatheter aortic valve implantation.

ELIGIBILITY:
Inclusion Criteria:

* Aged > 18 years
* Undergoing transfemoral TAVI with any commercially available transcatheter heart valve
* Provided written informed consent

Exclusion Criteria:

* Documented protamine allergy or anaphylaxis
* Recent PCI (< 3 months before TAVI)
* Planned arterial access via surgical cut-down

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Composite of all-cause mortality or type 1-4 bleeding | 30 days after TAVI
  According to the VARC-3 criteria

SECONDARY OUTCOMES:
All bleeding | 30 days after TAVI
  According to the VARC-3 criteria type 1-4 bleeding
Major, life-threatening or fatal bleeding | 30 days after TAVI
  According to the VARC-3 criteria type 2-4 bleeding
Major vascular complications | 30 days after TAVI
  According to the VARC-3 criteria
Cardiovascular mortality | 30 days after TAVI
  According to the VARC-3 criteria
All-cause mortality | 30 days after TAVI
  According to the VARC-3 criteria

OTHER OUTCOMES:
Safety endpoint: Anaphylaxis | 30 days after TAVI
  According to the National Institute of Allergy and Infectious Disease criteria
Safety endpoint: Thromboembolic events | 30 days after TAVI
  Composite of myocardial infarction, ischaemic stroke, transient ischaemic attack or non-cerebral distal embolization according to the VARC-3 criteria
Neurologic events | 30 days after TAVI
  According to the VARC-3 criteria
Hospitalization | 30 days after TAVI
  According to the VARC-3 criteria
Vascular and access-related complications | 30 days after TAVI
  According to the VARC-3 criteria
Cardiac structural complications | 30 days after TAVI
  According to the VARC-3 criteria
Other procedural or valve-related complications | 30 days after TAVI
  According to the VARC-3 criteria
New conduction disturbances and arrhythmias | 30 days after TAVI
  According to the VARC-3 criteria
Acute kidney injury | 30 days after TAVI
  According to the VARC-3 criteria
Myocardial infarction | 30 days after TAVI
  According to the VARC-3 criteria
Bioprosthetic valve dysfunction | 30 days after TAVI
  According to the VARC-3 criteria
Leaflet thickening and reduced motion | 30 days after TAVI
  According to the VARC-3 criteria
Clinically significant valve thrombosis | 30 days after TAVI
  According to the VARC-3 criteria
Time to hemostasis | 30 days after TAVI
  Is defined as elapsed time after sheath removal and first observed and confirmed arterial hemostasis.
Haemoglobin level | 30 days after TAVI
Need for transfusion | 30 days after TAVI
  Any bleeding requiring transfusion of 1 or more units of whole blood/RBC
Procedural haemostasis failure | 30 days after TAVI
  Procedural haemostasis failure is defined as failure to achieve haemostasis at the arteriotomy site within 20 minutes or leading to alternative treatment (e.g. fem-stop device, or adjunctive endovascular ballooning/stenting).
Delayed haemostasis failure | 30 days after TAVI
  The occurrence of bleeding requiring prolonged manual compression or alternative interventions (new pressure bandage, fem-stop device, endovascular or surgical repair) after initial haemostasis was achieved and patient is no longer in the catheterization laboratory.
Post-procedural length of stay | 30 days after TAVI
  Post-procedural length of stay will be measured in the time (days) from procedure to discharge.
Freedom from mortality | 30 days after TAVI
  According to the VARC-3 criteria
Successful access, delivery of the device, and retrieval of the delivery system | 30 days after TAVI
  According to the VARC-3 criteria
Correct positioning of a single prosthetic heart valve into the proper anatomical location | 30 days after TAVI
  According to the VARC-3 criteria
Freedom from surgery or intervention related to the device or to a major vascular or access-related, or cardiac structural complication | 30 days after TAVI
  According to the VARC-3 criteria
Technical success | 30 days after TAVI
  According to the VARC-3 criteria
Freedom from surgery or intervention related to the device or to a major vascular or access-related or cardiac structural complication | 30 days after TAVI
  According to the VARC-3 criteria
Intended performance of the valve (mean gradient <20 mmHg, peak velocity <3 m/s, Doppler velocity index ≥0.25, and less than moderate aortic regurgitation) | 30 days after TAVI
  According to the VARC-3 criteria
Freedom from all-cause mortality | 30 days after TAVI
  According to the VARC-3 criteria
Freedom from all stroke | 30 days after TAVI
  According to the VARC-3 criteria
Freedom from VARC type 2-4 bleeding | 30 days after TAVI
  According to the VARC-3 criteria
Freedom from major vascular, access-related, or cardiac structural complication | 30 days after TAVI
  According to the VARC-3 criteria
Freedom from acute kidney injury stage 3 or 4 | 30 days after TAVI
  According to the VARC-3 criteria
Freedom from moderate or severe aortic regurgitation | 30 days after TAVI
  According to the VARC-3 criteria
Freedom from new permanent pacemaker due to procedure-related conduction abnormalities | 30 days after TAVI
  According to the VARC-3 criteria
Freedom from surgery or intervention related to the device | 30 days after TAVI
  According to the VARC-3 criteria

CONTACTS AND LOCATIONS:
Locations (6):
- Belgium (2):
  - A.S.Z. Aalst, Aalst
  - University Hospitals Leuven, Leuven
- Netherlands (4):
  - Maastricht UMC, Maastricht, Limburg
  - Leiden University Medical Center, Leiden, South Holland
  - St. Antonius Hospital, Nieuwegein, Utrecht
  - Amsterdam University Medical Center, Amsterdam

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Overduin DC, van Ginkel DJ, Dubois C, Lesizza P, Broeze GM, Montero-Cabezas JM, Rosseel L, van der Kley F, van Nuland PJ, Smits TP, Hemelrijk KI, Aarts HM, Rensing BJWM, Timmers L, Swaans MJ, Sonker U, Veenstra L, van 't Hof AWJ, Peper J, Tijssen JGP, Delewi R, Vriesendorp PA, Ten Berg JM. Routine versus selective protamine administration to reduce bleeding after TAVI: Rationale and design of the POPular ACE TAVI trial. Am Heart J. 2026 Mar;293:107296. doi: 10.1016/j.ahj.2025.107296. Epub 2025 Oct 31. PMID 41177203